CLINICAL TRIAL: NCT02537873
Title: Phase I Drug Interaction and Self Administration Studies of Compounds for Cocaine Use Disorder
Brief Title: Drug Interaction and Self Administration Studies of Compounds for Cocaine Use Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HM20003768; 1U54DA038999 (NIH)
Record Dates: First submitted 2015-08-25; First posted 2015-09-02 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Cocaine Use Disorder
Keywords: Cocaine Use Disorder
MeSH Terms: interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Lorcaserin and Cocaine IV (Experimental): Lorcaserin 10 mg administered orally once daily for 6 days then increasing to twice daily for 3 days.
  Cocaine IV (intravenous) administered in ascending doses of 0, 10, 20, 40 mg on study days 1, 2, 6 and 12.
  Interventions: Drug: Lorcaserin; Drug: Cocaine Intravenous (IV)
- Arm 2: Placebo Comparator and Cocaine IV (Placebo Comparator): Dextrose placebo in gelatin capsule identical to experimental drug. Cocaine IV (intravenous) administered in ascending doses of 0, 10, 20, 40 mg on study days 1, 2, 6 and 12.
  Interventions: Drug: Cocaine Intravenous (IV); Drug: Placebo comparator

INTERVENTIONS:
Drug: Lorcaserin — Lorcaserin HCL 10mg tablets (Belviq, Arena Pharmaceuticals)
  Other Names: Belviq
  Arms: Arm 1: Lorcaserin and Cocaine IV
Drug: Cocaine Intravenous (IV) — Cocaine IV administered at doses of 10, 20 and 40 mg during 4 dosing sessions
Drug: Placebo comparator — Dextrose in gelatin capsule
  Arms: Arm 2: Placebo Comparator and Cocaine IV

SUMMARY:
The overall goal of this project is to develop initial human data on effects of novel compounds on safety (interactions with cocaine) and efficacy (subjective response to cocaine and self administration data) in non-treatment seeking cocaine use disorder subjects. The compound to be studied will be the 5-HT2CR agonist lorcaserin. Lorcaserin and other 5-HT2CR agonists have been shown to reduce cocaine self-administration and cue reactivity in rodents. In addition there is human safety data in non-cocaine using subjects for lorcaserin as it is currently FDA approved for obesity, and safety data from a cocaine interaction study in rodents , but there is no human cocaine interaction/PK data and no PD data to support potential dosages for phase II clinical trials.

DETAILED DESCRIPTION:
The overall goal of this project is to develop initial human data on effects of novel compounds on safety (interactions with cocaine) and efficacy (subjective response to cocaine and self-administration data) in non-treatment seeking cocaine use disorder subjects. This project will provide innovative data on effects of novel compounds on cocaine self-administration in addition to needed safety data on drug interactions with cocaine. This is a Phase I human drug interaction study examining the safety of concurrent administration of cocaine with novel compounds, and the effects of the novel compounds on subjective response to cocaine and cocaine self-administration in non-treatment seeking cocaine use disorder subjects. This data will provide important information for go/no-go decisions on phase II clinical trials using medications as a tool to enhance abstinence. The initial compound to be studied will be the 5-HT2CR agonist lorcaserin, which has been shown to reduce cocaine self-administration and cue reactivity in rodents. In addition there is human safety data in non-cocaine using subjects for lorcaserin as it is currently FDA approved for obesity, but there is no human cocaine interaction/PK data and no PD data to support potential dosages for phase II clinical trials.

This is a single center, double-blind, placebo-controlled, randomized, 1b/2a study. 18 of subjects are planned. Each subject will be administered a single dose of study drug three times, one week apart, consisting each time of various doses of active or placebo. Each subject will receive three of the four experimental treatments. Subjects will be assigned to the treatments in random order. Evaluations will be taken at baseline and 4 hours at each of the 3 study visits.

Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study. If subjects meet inclusion criteria, they will be admitted as hospital inpatients during the 14 study days to prevent drug and alcohol use and maintain complete monitoring for adverse events.

The following treatment regimens will be used:

Lorcaserin will be 10mg once daily increasing to 10mg twice daily. Placebo or Comparator - identical placebo capsules administered at the same time as lorcaserin.

Total duration of subject participation including eligibility screening (Study days -3 - 0), on-unit study days (Study days 1-14), and follow-up visits (Study days 16 and 20) will be three weeks. Total duration of the study is expected to be 18 months.

Detailed description of the in-hospital portion of study (Study days 1-14) is as follows:

After a screening cocaine infusion to determine safety, eligible subjects will be randomized to Group A -placebo only or Group B -placebo followed by an ascending dose of lorcaserin. Six subjects will be assigned to Group A (placebo) and 12 subjects will be assigned to Group B (active lorcaserin).

1. Days 1-2: All subjects will receive placebo on days 1-2 in a single blind fashion. Vital signs including heart rate, blood pressure and respiration rate will be obtained 15 minutes before and 15, 30 and 60 minutes after placebo administration. Days 1-2 will be single-blind placebo, whereas all remaining study days will be double-blind.
2. Days 3-9: On days 3-9, subject group A will receive one placebo pill twice daily, and group B will receive one placebo pill in the morning and one matching lorcaserin 10 mg pill in the evening, for a total dose of 10 mg daily. ECG with QTc will be performed daily. If the QTc is prolonged greater than 30ms over baseline lorcaserin dosage will be held.
3. Days 10-12: subjects in group B will have a blinded dosage increase to 10 mg of lorcaserin twice daily. Vital signs including heart rate, blood pressure and respiration rate will be obtained 15 minutes before and 15, 30 and 60 minutes after placebo/lorcaserin administration. ECG with QTc will be performed daily under the supervision of a study physician. If the QTc is prolonged greater than 30ms over baseline lorcaserin dosage will be held.
4. Day 13 subjects in group B will be administered 10mg of lorcaserin in the morning only, and subjects in group A will be administered matching placebo in the morning. Subjects will be discharged on day 14.
5. Cocaine Infusion Sessions (Days 1, 2, 6, and 12): All subjects will undergo an ascending dose intravenous cocaine administration after admission on day 1 to ensure safety of later cocaine studies.

To assess the safety and subjective effects of cocaine in the presence of lorcaserin, subjects will receive ascending doses of intravenous cocaine (10 mg, 20 mg, 40 mg), with each cocaine administration separated by one hour. In addition, 0 mg cocaine (saline) infusion will be randomly given after the first dose of cocaine in order to aid in blinding investigators and subjects to the order of drug administration. Infusions will be carried out at 9:00am, 10:00am, 11:00am and 12:00pm (Day 1), or at 1:00 p.m., 2:00 p.m., 3:00 p.m., and 4:00 p.m. (Days 2, 6, and 12).

ELIGIBILITY:
In order to participate in this study, subjects must:

1. Males and females between 18 and 59 years-of-age.
2. Understand the study procedures and provide written informed consent.
3. Meet current DSM-5 criteria for cocaine use disorder, at least moderate severity, and current DSM-IV diagnosis of cocaine dependence, but are not seeking treatment.
4. Currently using cocaine by smoking or intravenous route of administration as determined by self-report and have a positive urine drug screen for cocaine during screening.
5. Have vital signs as follows: resting pulse below 95 bpm, blood pressures below 140 mm Hg systolic and 90 mm Hg diastolic.
6. Have no clinically significant abnormalities in the judgment of the study physician in hematology and chemistry laboratory tests including liver function tests.
7. Have sinus rhythm with normal conduction (including QTcF less than 440 ms) by ECG.
8. Have no contraindications for study participation as determined by medical history and physical examination.
9. Be able to demonstrate an understanding of study procedures and follow instructions including behavioral laboratory testing.
10. No pregnant or nursing women will be permitted in the study, and women must either be unable to conceive (i.e., surgically sterilized, sterile, or postmenopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device with spermicide, or condoms). Men will be advised to use condoms. All females must provide negative pregnancy urine tests before study entry, at each visit during the study, and at the end of study participation.
11. Have hemoglobin/hematocrit values within normal limits based on age and gender.

In order to participate in the study, subjects must not:

1. Meet current DSM-5 diagnosis of any psychoactive substance use disorder other than cocaine, opiates, marijuana, or nicotine. Diagnosis of mild to moderate use disorder for alcohol will not be considered exclusionary.
2. Have a DSM-5 axis I psychiatric disorder other than substance use disorder including but not limited to Bipolar Disorder, Major Depressive Disorder, ADHD, or Schizophrenia or a neurological disorder requiring ongoing treatment and/or making study participation unsafe.
3. Have any previous medically adverse reaction to cocaine, including loss of consciousness, chest pain, or epileptic seizure.
4. Have any clinically significant medical disorder including cardiovascular (including hypertension), pulmonary, CNS, hepatic, or renal disorder.
5. Have a history of seizures (excluding childhood febrile seizures), or loss of consciousness for more than 20 minutes.
6. Have significant current suicidal or homicidal ideation or a history of suicide attempt within the past 6 months.
7. Have conditions of probation or parole requiring reports of drug use to officers of the court.
8. Have impending incarceration.
9. Have a positive HIV test by self-report or history.
10. Be pregnant or nursing or not using a reliable form of contraception if able to conceive. All females must provide negative pregnancy urine tests at screening, and daily after hospital admission.
11. Have any other illness, or condition, which in the opinion of the PI would preclude safe and/or successful completion of the study.
12. Have a positive breath alcohol test or urine drug screening positive for drugs of abuse with the exception of cocaine, opiates, cocaine metabolites, and marijuana.
13. Have a score greater than 5 on the Clinical Opiates Withdrawal Scale (COWS) on any screening, monitoring or hospital study visit.
14. Subjects who are allergic to lorcaserin.
15. Subjects who have taken any investigational drug within 90 days prior to baseline.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2015-07; Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick G Moeller, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Institute for Drug and Alcohol Studies, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 29 participants enrolled and passed screening. 4 withdrew or were terminated prior to randomization resulting in 25 randomized participants.
Groups:
- Arm 1: Lorcaserin and Cocaine IV: Test Lorcaserin 10 mg administered orally once daily for 6 days then increasing to twice daily for 3 days.
  Cocaine IV (intravenous) administered in ascending doses of 0, 10, 20, 40 mg on study days 1, 2, 6 and 12.
  Lorcaserin: Lorcaserin HCL 10mg tablets (Belviq, Arena Pharmaceuticals)
  Cocaine Intravenous (IV): Cocaine IV administered at doses of 10, 20 and 40 mg during 4 dosing sessions
Period: Overall Study
Arm/Group | Arm 1: Lorcaserin and Cocaine IV | Arm 2: Placebo Comparator and Cocaine IV
Started | 17 | 8
Completed | 9 | 4
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Lorcaserin and Cocaine IV: Lorcaserin 10 mg administered orally once daily for 6 days then increasing to twice daily for 3 days.
  Cocaine IV (intravenous) administered in ascending doses of 0, 10, 20, 40 mg on study days 1, 2, 6 and 12.
  Lorcaserin: Lorcaserin HCL 10mg tablets (Belviq, Arena Pharmaceuticals)
  Cocaine Intravenous (IV): Cocaine IV administered at doses of 10, 20 and 40 mg during 4 dosing sessions
- Total: Total of all reporting groups
Arm/Group | Arm 1: Lorcaserin and Cocaine IV | Arm 2: Placebo Comparator and Cocaine IV | Total
Number analyzed (Participants) | 9 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.78 (5.29) | 56.25 (2.06) | 50.85 (6.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 8 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 3 | 11
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) - Heart Rate
Description: Change in Heart rate (HR) measures during saline infusions will be compared to HR and BP after each cocaine infusion.
Time Frame: Baseline to up to 5 hours on up to day 12 of the study
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Arm 1: Lorcaserin and Cocaine IV | Arm 2: Placebo Comparator and Cocaine IV
Number analyzed (Participants) | 9 | 4
beats per minute | 7.8 (7.98) | 4.96 (6.94)

2. Primary Outcome: Cocaine Self-administration Choice Selection
Description: During a study visit 13 days after participant enrollment, participants will be allowed to choose to receive an infusion of cocaine or $5. Number of times participants self-administered Cocaine over an approximately 2 1/2 hour period in the morning and in the afternoon will be counted.
Time Frame: 13 days
Measure: Mean (Standard Deviation); unit: cocaine infusions
Arm/Group | Arm 1: Lorcaserin and Cocaine IV | Arm 2: Placebo Comparator and Cocaine IV
Number analyzed (Participants) | 9 | 4
cocaine infusions
  morning self-administration | 2.125 (2.03) | 2.2 (2.28)
  afternoon self-administration | 0.4 (0.89) | 4.66 (0.81)

3. Primary Outcome: Change in Subjective Experience
Description: During a study visit, participants will be given an infusion of cocaine. Participants will rate their subjective craving for cocaine on a visual analog scale. The scale is rated from Not at all to Extremely. Scores are calculated by measuring in centimeters from Not at all (0) to where the participant marked with the highest score being 100. Participants will rate their subjective experience at baseline (prior to drug infusion) and after cocaine infusion.
Time Frame: Day 12, pre-infusion to post-infusion (up to 5 hours)
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Arm 1: Lorcaserin and Cocaine IV | Arm 2: Placebo Comparator and Cocaine IV
Number analyzed (Participants) | 9 | 4
Centimeters | 1.4 (8.5) | 1.33 (1.52)

4. Primary Outcome: Cocaine PK With Placebo
Description: Regardless of randomization category, all participants will receive the placebo on days 1 and 2 in a single blind fashion. Plasma concentration-time profiles of cocaine after cocaine infusion during placebo administration (Day 2) will be analyzed to determine how many participant's pharmacokinetic (PK) parameter estimates after using cocaine differ from expected PK parameter estimates for a typical individual using cocaine.
Time Frame: 2 days
Measure: Number; unit: participants
Arm/Group | Arm 1: Lorcaserin and Cocaine IV | Arm 2: Placebo Comparator and Cocaine IV
Number analyzed (Participants) | 9 | 4
participants | 0 | 0

5. Primary Outcome: Cocaine PK With Study Drug
Description: Plasma concentration-time profiles of cocaine after cocaine infusion during study drug (Lorcaserin or placebo) administration (Day 12) will be analyzed to determine how many participant's pharmacokinetic (PK) parameter estimates after using cocaine differ from expected PK parameter estimates for a typical individual using cocaine.
Time Frame: Day 12
Measure: Number; unit: participants
Arm/Group | Arm 1: Lorcaserin and Cocaine IV | Arm 2: Placebo Comparator and Cocaine IV
Number analyzed (Participants) | 9 | 4
participants | 0 | 0

6. Secondary Outcome: Response Inhibition During Immediate Memory Task (IMT)
Description: Commission errors on the IMT (Immediate Memory Task) will be compared between lorcaserin and placebo subjects to determine the extent to which this measure is modified by the administration of lorcaserin using repeated measures ANOVA.
Time Frame: 3 days (Study days 1, 8, 11)
Population: Data was not collected
Arm/Group | Arm 1: Lorcaserin and Cocaine IV | Arm 2: Placebo Comparator and Cocaine IV
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) - Change in Blood Pressure
Description: Change in blood pressure (BP) measures during saline infusions will be compared to HR and BP after each cocaine infusion.
Time Frame: Day 12, baseline to final cocaine infusion (approximately 5 hours)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Arm 1: Lorcaserin and Cocaine IV | Arm 2: Placebo Comparator and Cocaine IV
Number analyzed (Participants) | 9 | 4
mmHg
  Systolic Blood Pressure (BP) | 6.2 (4.55) | 4.27 (11.28)
  Diastolic BP | 0.4 (6.65) | 3.54 (4.79)

ADVERSE EVENTS:
Time Frame: 19 days - from 1st study visit to final follow-up.
Description: Adverse Events (AEs) will be identified through daily interviews with participants and noted at any visit.
Arm/Group | Arm 1: Lorcaserin and Cocaine IV | Arm 2: Placebo Comparator and Cocaine IV
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/4
Other Adverse Events (participants affected / at risk) | 2/9 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Lorcaserin and Cocaine IV (N=9) | Arm 2: Placebo Comparator and Cocaine IV (N=4)
QTc prolongation (Cardiac disorders) | 1 (1) | 0 (0)
chest tightness (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT02537873/Prot_SAP_000.pdf